CLINICAL TRIAL: NCT04565002
Title: Effect of Transcutaneous Electrical Diaphragmatic Stimulation on Respiratory Muscle Strength, Diaphragm Thickness and Mechanical Ventilation Time in Critically Ill Elderly Patients
Brief Title: Transcutaneous Electrical Diaphragmatic Stimulation in Critically Ill Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2020-09-18; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: ICU Acquired Weakness; Diaphragmatic Injury
Keywords: transcutaneous electrical diaphragmatic stimulation; elderly; mechanical ventilation; ICU acquired weakness

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: The study has a double blind characteristic. Neither the researcher nor the research subject is aware of his group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EG (Experimental): The TEDS protocol will consist of the following parameters: a) frequency of 30 Hz; b) pulse width of 0.4 ms; c) respiratory rate of 15 irpm; d) holding time of 1 s; e) rise time of 1 s; f) 2 s descent time; and g) 2 s non-stimulus time. Phrenics equipment (Dualpex 961, Quark®) will be used. The positioning of the electrodes will be performed according to a study by Cancelliero et al. (2012), who proposed the placement of two electrodes in the right and left paraxiphoid regions, and two others in the direction of the axillary midline, over the seventh intercostal space, also on the right and left sides.
  Interventions: Device: Transcutaneous Electrical Diaphragmatic Stimulation
- CG (No Intervention): The control group will undergo the same assessments as the experimental group, but the TEDS will not be applied.

INTERVENTIONS:
Device: Transcutaneous Electrical Diaphragmatic Stimulation — The procedure consists of electrical stimulation in the region of the motor points of the diaphragm. Its configurations contribute to produce involuntary muscle contractions. There are four electrodes positioned superficially on the skin.
  Other Names: TEDS
  Arms: EG

SUMMARY:
Abstract..........................................................................................................04 Introduction....................................................................................................10 Methods.........................................................................................................14 Financial Support...........................................................................................22 References.....................................................................................................24

DETAILED DESCRIPTION:
1. INTRODUCTION Patients undergoing invasive mechanical ventilation (IMV) have an intense predisposition to the development of muscle weakness in the first hours after the orotracheal intubation process, since they are exposed, among other factors, to sedative drugs, immobilization and properly controlled ventilation (DEMOULE et al., 2016). It is observed that approximately 25% to 50% of patients submitted to ventilatory support have muscle weakness and, of this proportion, 85% to 95% persist with neuromuscular impairment for a period of two to five years.

   In this context, the elderly deserve attention because the demographic transition process has the inversion of the age pyramid as one of its characteristics (WONG et al., 2006). This leads to a higher incidence of admissions of these patients in intensive care units compared to young people and adults, considering that they represent the largest portion of the population.

   Among the muscles affected by permanence in IMV in the general population and especially in the elderly, the diaphragm can be highlighted, which evolves with a reduction in its ability to generate tension due to the atrophy of its muscle fibers. This leads to an alteration called diaphragmatic dysfunction (DD). The mechanisms involved with DD are the reduction in the number of myofibrils (proteins that involve filaments of actin and myosin responsible for the production of muscle contraction), oxidative stress (inducing the activation of the forkhead box O1 protein, involved with the processes of gluconeogenesis and glycogenolysis) and the abnormal activation of a pathway responsible for the proteolysis of adenosine triphosphate, ubiquitin-proteasome.

   Considering the progressive characteristic of DD, some consequences such as increased IMV time, increased risk of respiratory complications and prolonged hospital stay can be observed, if no specific intervention is performed . Therefore, it is necessary to adopt measures that allow the early detection of diaphragmatic weakness, as well as the use of conducts that prevent or treat this clinical condition.

   As for the diagnosis of DD, it can be performed using instruments that measure inspiratory muscle strength, such as the manovacuometer, in addition to imaging tests that show the diaphragmatic thickness (FDI), such as pulmonary ultrasonography (PU) . The variable referring to inspiratory muscle strength in manovacuometry is the maximum inspiratory pressure (MIP), while the thickness of the diaphragm, verified through the PU, is represented by the diaphragmatic thickening index (DTI), obtained through the difference between the diaphragm thickness total lung capacity (DTTLC) and functional residual capacity (DTFRC), divided by DTTLC. The FDI contributes to the initial diagnosis of DD and is also relevant for monitoring the evolution of diaphragm function during the period of hospitalization and ventilatory weaning. According to Goligher et al. (2015), the decrease in FDI is associated with impaired function of the diaphragm and is correlated with low values of MIP in critically ill patients.

   After obtaining variables related to the function of the diaphragm, as previously described, conducts aimed at preventing or treating DD are important in an attempt to minimize possible damage to the critical patient. Within outpatient pulmonary rehabilitation, positive effects have been demonstrated with the use of electrotherapy, specifically through the technique of transcutaneous electrical diaphragmatic stimulation (TEDS) in patients with chronic obstructive pulmonary disease (COPD). This technique consists of placing electrodes on the skin, in places close to the motor points of the diaphragm, transmitting an intermittent current and generating action potentials capable of producing muscle contractions. However, in the literature, there is no evidence on the effects of this therapy on the FDI of elderly critically ill patients, or even to assess the impact of TEDS on the time of mechanical ventilation and hospitalization of this population. In view of the practicality of this treatment, its low cost and the scarcity of evidence on this topic, the objective of the present study will be to assess the influence of TEDS on respiratory muscle strength, diaphragm thickness and duration of mechanical ventilation in critically ill patients under care intensive.
2. METHODS

   2.1. Study Design and Recruitment

   The present study will be a controlled randomized clinical trial. It will also be registered in the Clinical Trials.

   All research participants will be submitted to the assessment of respiratory muscle strength (manovacuometry) and diaphragm thickness (PU), and only EG patients will be exposed to an intervention through the use of TEDS.

   2.2. Sample

   The sample will consist of participants of both sexes, over the age of 60, who have undergone IMV. The research participants will be divided into a control group (CG) and an experimental group (EG) and will carry out the same evaluation steps during the spontaneous breathing test after weaning from mechanical ventilation, with only the EG undergoing TEDS. The details of the intervention will be exposed later.

   2.3 Proposed Procedures / Methods

   The evaluation of the research subjects will take place in the Adult Intensive Care Units (I and II) of the Hospital e Maternidade Therezinha de Jesus - Juiz de Fora.

   2.3.1. Distribution of Participants, Evaluation and Intervention

   The research participants will be submitted to the evaluation of the FDI through the PU, as well as of the respiratory muscle strength, through the manovacuometry, immediately after the ventilatory weaning. It is worth noting that weaning and extubation will be carried out following an institutional checklist (Appendix I) for greater patient safety.

   The EG, immediately after the 24-hour period on VMI, will be submitted to TEDS, twice a day, with an interval of six hours between therapies to prevent respiratory muscle fatigue. Initially, it will be performed with the patient in assisted-controlled ventilation mode and well adapted to ventilation. The sensitivity parameter will be adjusted to the value necessary so that the contractions produced by electrical stimulation do not trigger the mechanical ventilator, preventing episodes of asynchrony. After the suspension of drugs with a sedative effect (such as benzodiazepines and endogenous opioids) and the ventilatory drive is resumed, TEDS will continue to be used in EG patients until extubation, in spontaneous ventilation, following the same protocol, however with the sensitivity readjusted to the standardized values to prevent muscle fatigue. The procedures will be detailed below.

   2.3.2. Pulmonary Ultrasound

   Ultrasonography is a simple, safe and relatively low-cost procedure that, when using exact equipment and standardized techniques applied by trained professionals, provides relevant information on the respiratory system that has been demonstrated over the last few years (DEMI et al., 2014).

   The patient will position himself in the supine position and there will be the use of the linear transducer to evaluate the superficial structures and the cardiac transducer to evaluate the deep ones. There is a wide range of techniques to be employed, but the eight-zone assessment is practical and quick to perform in emergency assessment and in intensive care patients. The latter consists of the scanning of four areas by hemithorax, namely: zones 1 and 2 indicate the upper anterior chest wall and the lower anterior one respectively, and zones 3 and 4 indicate the upper lateral chest wall as well as the lower lateral wall, respectively.

   The equipment used to perform all pulmonary ultrasound exams will be the GE LogiqE (Logiq-E GE 2014, Contagem, MG, Brazil), from the Ultrasonography Sector of the Hospital and Maternidade Terezinha de Jesus, Juiz de Fora (MG).

   2.3.3. Assessment of Respiratory Muscle Strength

   According to the American Thoracic Society (2002), the appropriate protocol for obtaining the measurements related to respiratory muscle strength (MIP) must respect the following characteristics: a) environment with a temperature of approximately 21ºC; b) previous calibration of the manovacuometer; c) patient in a sitting posture (head elevated by 90 °); and d) execution of a maximum inspiration starting from the residual volume (RV) to reach the total lung capacity (TLC). The procedure must be repeated two more times, with an interval of two minutes between repetitions (prevention of muscle fatigue) and the measures of MIP and maximum expiratory pressure (MEP) considered will be the highest recorded. The equipment used will be brand M120, with a scale of 4 cmH2O, with variation of +/- 120 cmH2O.

   2.3.4. Transcutaneous Electrical Diaphragmatic Stimulation

   The TEDS protocol will consist of the following parameters: a) frequency of 30 Hz; b) pulse width of 0.4 ms; c) respiratory rate of 15 irpm; d) holding time of 1 s; e) rise time of 1 s; f) 2 s descent time; and g) 2 s non-stimulus time. Phrenics equipment (Dualpex 961, Quark®, SP, Brazil) will be used. The positioning of the electrodes will be performed according to a study by Cancelliero et al. (2012), who proposed the placement of two electrodes in the right and left paraxiphoid regions, and two others in the direction of the axillary midline, over the seventh intercostal space, also on the right and left sides. The duration of the procedure will be 30 minutes, twice a day, with a six-hour interval between applications, until the patient undergoes the extubation process. As long as it does not have a level of consciousness, is not in spontaneous ventilatory mode and without the use of drugs with a sedative effect, the sensitivity of the ventilator will be adjusted in a way that does not trigger the equipment, to avoid episodes of asynchrony. Immediately after recovering the level of consciousness, resuming the ventilatory drive and suspending sedative drugs, the patient during TEDS will be stimulated to inhale after the perception of the arrival of the electric current, in spontaneous mode, and with the sensitivity adjusted to the baseline values.

   2.3.4. Scratchs

   There are chances of hemodynamic decompensation and respiratory distress during the use of TEDS in EG patients, including changes in heart rate, blood pressure, as well as respiratory rate and synchronization with the mechanical ventilator. If the events described occur, the TEDS procedure will be stopped immediately. Ventilatory adjustments will be made by the researcher according to the demands presented and the doctor on duty will be informed to adopt conducts aimed at the patients' hemodynamic recovery, regarding medication adjustments. There will be supervision by the responsible researcher and the rest of the multidisciplinary team.

   2.3.5. Benefits

   Benefits may be generated for the study participants, including the reduction in the time of mechanical ventilation, hospitalization, in addition to the probable rapid reintegration of patients into activities of daily living after discharge, since diaphragmatic muscle weakness contributes substantially to the delay in the process of recovering functionality.
3. FINANCIAL SUPPORT

The equipment used in the research is available at the Therezinha de Jesus Hospital and Maternity Hospital in the city of Juiz de Fora, state of Minas Gerais.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 60 years who underwent IMV.

Exclusion Criteria:

* Recent surgical scar and/or open lesion in the regions where the electrodes would be placed
* Severe hemodynamic instability
* Patient-ventilator asynchrony not reversible with adjustments or optimization of sedation
* Hypoglycemia < 60 mg/dL
* Presence of a cardiac pacemaker
* Undrained pneumothorax
* Use of increasing doses of vasoactive drugs.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
As a primary endpoint, the change in FDI in EG patients will be considered. | 18 months
  This index is considered valid to predict success in weaning and extubation, together with other variables.

SECONDARY OUTCOMES:
Changes in mechanical ventilation time | 20 months
  The change in mechanical ventilation time may favor hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital e Maternidade Therezinha de Jesus, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sassoon CS, Caiozzo VJ, Manka A, Sieck GC. Altered diaphragm contractile properties with controlled mechanical ventilation. J Appl Physiol (1985). 2002 Jun;92(6):2585-95. doi: 10.1152/japplphysiol.01213.2001. PMID 12015377
- [Result] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Result] Delerme S, Ray P. Acute respiratory failure in the elderly: diagnosis and prognosis. Age Ageing. 2008 May;37(3):251-7. doi: 10.1093/ageing/afn060. Epub 2008 Apr 3. PMID 18388161
- [Result] Demoule A, Molinari N, Jung B, Prodanovic H, Chanques G, Matecki S, Mayaux J, Similowski T, Jaber S. Patterns of diaphragm function in critically ill patients receiving prolonged mechanical ventilation: a prospective longitudinal study. Ann Intensive Care. 2016 Dec;6(1):75. doi: 10.1186/s13613-016-0179-8. Epub 2016 Aug 5. PMID 27492005
- [Result] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Result] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Result] Gargani L, Volpicelli G. How I do it: lung ultrasound. Cardiovasc Ultrasound. 2014 Jul 4;12:25. doi: 10.1186/1476-7120-12-25. PMID 24993976
- [Result] Geddes LA, Voorhees WD, Bourland JD, Riscili CE. Optimum stimulus frequency for contracting the inspiratory muscles with chest-surface electrodes to produce artificial respiration. Ann Biomed Eng. 1990;18(1):103-8. doi: 10.1007/BF02368420. PMID 2306029
- [Result] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Result] Hussain SN, Mofarrahi M, Sigala I, Kim HC, Vassilakopoulos T, Maltais F, Bellenis I, Chaturvedi R, Gottfried SB, Metrakos P, Danialou G, Matecki S, Jaber S, Petrof BJ, Goldberg P. Mechanical ventilation-induced diaphragm disuse in humans triggers autophagy. Am J Respir Crit Care Med. 2010 Dec 1;182(11):1377-86. doi: 10.1164/rccm.201002-0234OC. Epub 2010 Jul 16. PMID 20639440
- [Result] Kim WY, Lim CM. Ventilator-Induced Diaphragmatic Dysfunction: Diagnosis and Role of Pharmacological Agents. Respir Care. 2017 Nov;62(11):1485-1491. doi: 10.4187/respcare.05622. Epub 2017 Jul 11. PMID 28698263
- [Result] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Result] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Result] Radell PJ, Remahl S, Nichols DG, Eriksson LI. Effects of prolonged mechanical ventilation and inactivity on piglet diaphragm function. Intensive Care Med. 2002 Mar;28(3):358-64. doi: 10.1007/s00134-002-1207-8. Epub 2002 Feb 6. PMID 11904668
- [Result] Umbrello M, Formenti P, Longhi D, Galimberti A, Piva I, Pezzi A, Mistraletti G, Marini JJ, Iapichino G. Diaphragm ultrasound as indicator of respiratory effort in critically ill patients undergoing assisted mechanical ventilation: a pilot clinical study. Crit Care. 2015 Apr 13;19(1):161. doi: 10.1186/s13054-015-0894-9. PMID 25886857
- [Result] van den Berg M, Hooijman PE, Beishuizen A, de Waard MC, Paul MA, Hartemink KJ, van Hees HWH, Lawlor MW, Brocca L, Bottinelli R, Pellegrino MA, Stienen GJM, Heunks LMA, Wust RCI, Ottenheijm CAC. Diaphragm Atrophy and Weakness in the Absence of Mitochondrial Dysfunction in the Critically Ill. Am J Respir Crit Care Med. 2017 Dec 15;196(12):1544-1558. doi: 10.1164/rccm.201703-0501OC. PMID 28787181
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837